CLINICAL TRIAL: NCT04138628
Title: Treatment Of Metastatic Bladder Cancer at the Time Of Biochemical reLApse Following Radical Cystectomy
Acronym: TOMBOLA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jørgen Bjerggaard Jensen (Other)
Collaborators: Aarhus University Hospital (Other); Herlev Hospital (Other); Rigshospitalet, Denmark (Other); Odense University Hospital (Other); Aalborg University Hospital (Other)
Responsible Party: Sponsor-Investigator, Jørgen Bjerggaard Jensen, MD, DMSc, Professor, Consultant in Urology, Aarhus University Hospital
Organization: Aarhus University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DaBlaCa-14; 2019-001679-36 (EudraCT Number)
Record Dates: First submitted 2019-10-23; First posted 2019-10-24 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Bladder Cancer; Bladder Cancer, Metastatic
Keywords: Muscle Invasive Bladder Cancer (MIBC); biomarkers; ctDNA; immunotherapy; circulating tumor DNA; liquid biopsies
MeSH Terms: conditions — Urinary Bladder Neoplasms; Neoplasm Metastasis | interventions — atezolizumab

STUDY DESIGN:
Intervention Model Description: Single country Investigator Initiated, Open-label, Single-arm, Non-randomized, Phase II study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ctDNA screening arm (Experimental): Flat dose 1200 mg Atezolizumab every three weeks for up to 13 months
  Interventions: Drug: Atezolizumab

INTERVENTIONS:
Drug: Atezolizumab — The study drug will be given according to current recommendations as systemic treatment every third week for 12 months or until progression. Treatment will be initiated within 28 days of detection of ctDNA.

SUMMARY:
Immunotherapy (checkpoint inhibitors) is approved as first and second line treatment to patients with metastatic bladder cancer. However, response rates are low and no biomarkers have yet shown strong predictive value for patient selection. Moreover, the term 'metastatic' is based on metastases visible on conventional CT scans and, thus, require a certain size of tumour load. Clinical trials are currently being conducted that investigate the use of adjuvant immunotherapy for this group of patients (treatment to all), which will result in massive over-treatment and huge costs to the healthcare system.

This project has the primary objective to identify new indications for initiating immunotherapy in patients with metastatic bladder cancer. Sensitive molecular techniques for detection of tumor DNA in the blood will be used to identify patients with early signs of metastatic disease. In addition, comprehensive biomarker analysis will be performed to identify predictors of treatment response.

DETAILED DESCRIPTION:
The study aim at investigate the response rate and oncological outcome of systemic immunotherapy (PDL-1 inhibitor; atezolizumab) administered early at the time of biochemical relapse (circulating tumor DNA (ctDNA) positive) in patients who have undergone radical cystectomy because of muscle invasive bladder cancer.

Biomarkers that predict response to systemic immunotherapy will be identified by comprehensive multi-omics analysis of primary tumors and metastatic lesions. Furthermore, we will determine if ctDNA levels during therapy can be used as a biomarker for early indication of therapy response.

The hypotheses is that 1) early initiation of immunotherapy in high-risk (ctDNA positive) patients will result in better response rates and improved survival compared to later treatment following conventional imaging diagnosis of metastasis, and 2) biomarkers for predicting response can be identified and used for tailoring treatment regimens in the future to patients at high risk and at high likelihood of response.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age at the time of signing the Informed Consent Form
* For male study subjects: agreement to remain abstinent (refrain from heterosexual intercourse) or use a condom, and agreement to refrain from donating sperm.
* Signed Informed Consent Form
* ECOG PS 0, 1 or 2
* Is, according to the Investigator's judgement, able to comply with the trial protocol
* Ability to understand the Participant Information Sheet orally and in writing
* Preoperative PET/CT of thorax, abdomen, and pelvis with no suspicion of organ metastases or lymph node metastasis* above the aortic bifuraction
* Study Subjects undergoing radical cystectomy due to histologically documented muscle invasive urothelial carcinoma (including subtypes) stage cT2-4a in the urinary bladder following NAC** in cisplatin-fit Study Subjects.

  * Study Subjects who have undergone down-staging chemotherapy because of lymph node metastasis with no organ metastases can be included if complete response regarding lymph nodes are identified on preoperative imaging.

    * NAC includes Study Subjects who have stopped after one course of chemotherapy because of side effects or local non-metastatic progression

Exclusion Criteria:

* Subjects undergoing non-radical cystectomy for palliative reasons
* Non-radical surgery estimated intraoperative
* Other histology of BC than urothelial carcinoma - mixed tumours with urothelial features are allowed
* Concomitant invasive cancer within 5 years other than non-melanoma skin cancer and prostate cancer without metastasis
* Known contraindication to immunotherapy
* A history of autoimmune disease. Study Subjects with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll. Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
* Study Subjects who meet any of the following criteria will be excluded from study entry:

  * History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan
  * Treatment with systemic immunostimulatory agents (including, but not limited to, interferon and interleukin 2 [IL-2]) within 4 weeks or 5 drug elimination half-lives (whichever is longer) prior to initiation of study treatment
* HIV positive
* History of pneumonitis (History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
* Hepatitis B or hepatitis C infection
* Subjects who have received a live, attenuated vaccine within 28 days prior to enrolment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Estimated)
Dates: Start 2020-03-24 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2029-11-01 (Estimated)

PRIMARY OUTCOMES:
Complete response (CR) after treatment with investigational agent initiated by ctDNA positive status after radical cystectomy (with or without concomitant visible metastases on CT). | Time from treatment initiation with investigational agent until 12 months after initiation
  CR in the current study is defined as ctDNA negative status combined with regular imaging (CT) after treatment. Thus, any metastasis visible on CT at the time of treatment initiation should undergo complete response. In Study Subjects without visible metastasis on CT at the time of treatment, initiation should result in unchanged status on CT.
  Data will be compared to available historical data on response to PD-1 / PD-L1 targeted agents.

SECONDARY OUTCOMES:
Duration of freedom from clinical relapse in Study Subjects showing decrease or stabilization of ctDNA level after treatment with investigational agent | 12 months
  Time from initiation of therapy until response
Overall survival after cystectomy in Study Subjects having biochemical relapse | 5 years
  Percentage
Cancer specific survival after cystectomy in Study Subjects having biochemical relapse | 5 years
  Percentage
Recurrence free survival after cystectomy in Study Subjects having biochemical relapse | 5 years
  Percentage
Cancer specific survival after cystectomy in Study Subjects having biochemical relapse stratified for potential predictive biomarkers for response to treatment | 5 years
  Percentage
Response rate to investigated agent stratified for PD-L1 expression and other predictive biomarkers like TMB, immune cell infiltration, tumor subtypes etc. | 12 months
  Percentage
Time to recurrence seen on imaging (symptomatic or asymptomatic) | 5 years
  Percentage

CONTACTS AND LOCATIONS:
Overall Officials: Jørgen B Jensen, Professor, Principal Investigator — Dept. Of Urology, Aarhus University Hospital, Denmark; Lars Dyrskjøt, Professor, Study Chair — Dept. Of Molecular Medicine (MOMA) Aarhus University Hospital, Denmark; Mads Agerbæk, MD, Principal Investigator — Dept. Of Oncology, Aarhus University Hospital, Denmark; Karin Birkenkamp-Demtröder, Ass. professor, Study Chair — Dept. Of Molecular Medicine (MOMA) Aarhus University Hospital, Denmark
Locations (5):
- Denmark (5):
  - Aalborg Universitetshospital, Aalborg
  - Aarhus University Hospital, Aarhus
  - Rigshospitalet, Copenhagen
  - Herlev Hospital, Herlev
  - Odense Universitetshospital, Odense

IPD SHARING:
Plan to Share IPD: No